CLINICAL TRIAL: NCT04630834
Title: Oral Ibuprofen Plus Acetaminophen Versus Ibuprofen Alone for Acute Pain Reduction in Children
Brief Title: Ibuprofen Plus Acetaminophen for Enhanced Pain Reduction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Sandra Cunningham, MD, Division Director, Pediatric Emergency Medicine, New York City Health and Hospitals Corporation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-12329
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute
Keywords: children
MeSH Terms: conditions — Acute Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Two arms will be run in parallel. One arm will be acetaminophen and ibuprofen combined. The other arm will be ibuprofen alone with a placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Intervention Group: ibuprofen 10 mg/kg (maximum 600mg) plus acetaminophen 15mg/kg (maximum 650mg)
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen
- Placebo Group (Placebo Comparator): Placebo Group: Ibuprofen 10mg/kg (maximum 600 mg) plus placebo 15mg/kg (maximum 650mg)
  Interventions: Drug: Ibuprofen; Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Patients will receive both ibuprofen 10mg/kg weight based dosing with a max of 600mg
Drug: Acetaminophen — patients will receive acetaminophen 15 mg/kg weight based dosing with a max of 650mg
  Arms: Intervention group
Drug: Placebo — patients will receive placebo 15mg/kg weight based dosing with a max of 650mg
  Arms: Placebo Group

SUMMARY:
Combination of analgesics with different modes of action have the potential to offer enhanced pain relief with reduced dosage. Ibuprofen and acetaminophen have different modes of action. Combination of ibuprofen and acetaminophen has shown enhanced analgesia in adult studies, with pediatric data limited to post-operative pain and dental pain. Our study objective is to evaluate the analgesic efficacy of oral acetaminophen plus ibuprofen versus ibuprofen plus placebo for the management of acute pain in a pediatric emergency department.

DETAILED DESCRIPTION:
In the pediatric emergency department (PED), acute traumatic and nontraumatic pain accounts for approximately 9% of ED visits. The initial drugs of choice for analgesia are typically ibuprofen or acetaminophen. Both drugs display analgesic and antipyretic effects via distinct mechanisms of action. Various meta-analyses in the literature have compared ibuprofen and acetaminophen for pain relief in adults and children. Ibuprofen has been shown to be very effective for mild to moderate pain, especially in musculoskeletal injuries, including some limb fractures.

Combination of analgesics with different modes of action have the potential to offer enhanced pain relief with reduced dosage. Ibuprofen and acetaminophen have different modes of action. Ibuprofen is an NSAID that inhibits the activity of cyclooxygenase-1 and cyclooxygenase-2 enzymes and blocks the synthesis of prostaglandins and thromboxanes. The mode of action of acetaminophen for its analgesic effects is not entirely understood. It is thought that its effects are mediated through serotonergic pathways, cannabinoid and nitric oxide synthase, substance P, and N-methyl-D-aspartate. Combination of ibuprofen and acetaminophen has shown enhanced analgesia in adult studies, with pediatric data limited to post-operative pain and dental pain.

The data is limited regarding the combination of acetaminophen and ibuprofen for acute pain in the PED. A recent study showed similar analgesic efficacy of oral ibuprofen and acetaminophen in comparison with each analgesic alone for short-term treatment of acute pain in the PED7. In this study, pain reassessment was limited to only one time point at 60 minutes and included patients with pain scores of 1 on a 10 point scale. Since there is ample data demonstrating the effectiveness of ibuprofen for pain, we will investigate whether the combination of ibuprofen plus acetaminophen is superior for moderate to severe pain reduction compared to ibuprofen alone.

Objective To evaluate the analgesic efficacy of oral acetaminophen plus ibuprofen versus ibuprofen plus placeboalone for the management of acute pain in a pediatric emergency department.

Hypothesis: The combination of oral acetaminophen and ibuprofen is superior to ibuprofen alone for the reduction of acute traumatic and nontraumatic pain.

Study Design This will be a prospective, double-blind, placebo-controlled randomized trial, conducted in the pediatric emergency department.

Participant Recruitment Patients ages 3 years through 20 years who present to the PED with traumatic and/or nontraumatic pain will be assessed for eligibility. Pain assessment will be performed by a study investigator upon presentation at triage before medication administration. A validated numeric pain score (11-point 0-10 scale) will be used for patients 8 through 20 years. The Wong-Baker FACES Pain Scale (11-point 0-10 scale) will be used for patients ages 3 through 7 years. If the patient is eligible for enrollment, details of the study will be discussed with parent and/or patient and consent/assent will be obtained if they agree to participate.

Female patients >12 years will be assessed for pregnancy with a point of care urine HCG test. Pregnant patients will be excluded. Patients found to be pregnant will not be enrolled in the study and will be given appropriate care as is our standard procedure.

Study Intervention Study participants will be randomized to one of two treatment groups according to predetermined block randomization. A clinical research pharmacist will prepare placebo and acetaminophen in identical 20 mL amber bottles labeled sequentially. The bottle, 5, 10 and 20 mL amber syringes, and study documents will be stored in individual sequentially numbered manilla envelopes in a locked cabinet in the PED medication room. A nurse will draw the appropriate weight-based dose of placebo or medication into the amber syringes and administer the placebo or medication to the patient. Additionally, the nurse will administer a weight based dose of ibuprofen to each study participant.

The placebo group will receive a single weight-based dose of oral ibuprofen (100mg/5mL) at 10mg/kg to a maximum of 600 mg and placebo, mirrored as acetaminophen concentration of 160mg/5mL, at 15mg/kg to a maximum of 20 mL. The intervention group will receive a weight-based dose of ibuprofen (100mg/5mL) at 10mg/kg to a maximum of 600 mg and a dose of acetaminophen (160mg/5mL) at 15mg/kg to a maximum of 20 mL (650mg). The patient will then be evaluated in a standard manner by a treating clinician. The study investigator will reassess the pain score at 1 hour and 2 hours after medication administration. At the discretion of the treating physician, patients will receive parenteral medications at any time during the two hour assessment period for increasing or unremitting pain. Patients who are ready for discharge before the two hour pain assessment will receive a final pain score by the study investigator with documentation of time of the reassessment. Adverse events during the assessment period will be documented on a data collection sheet.

Subject treatment assignments will remain blinded until the final subject has completed follow up and all data has been recorded and validated. Urgent, immediate unblinding due to medical emergency may be authorized by the Investigator. When possible, the treatment assignment will be provided to the treating physician in order to maintain the blind for the Investigator and study staff. All instances of subject unblinding will be documented in the study record

Consent Written informed consent will be obtained by a study investigator at triage before initiation of treatment. An informed consent will be obtained parent or legal guardian for all patients 17 years and younger. Patients ages 13 years and older will sign an informed consent and an assent will be obtained from patients 7 years to 12 years of age.

Patients who are in pain and are first approached at the time the protocol will be initiated must be capable of providing contemporaneous informed consent. The principal investigator or study investigator will assess the capacity of the patient to provide ethically adequate informed consent. If the patient has capacity and consents to participation these facts will be documented in the patient's research record.

Confidentiality All patient data and research records will be kept confidential. Data collection sheets will be stored in a locked cabinet in the principal investigator's locked office throughout the study period and will be accessible only to research staff. Data will be collected on paper forms then entered into a password protected computer database. After data collection is performed, identifiers will be removed from the data file. Research investigators responsible for study collection, nurses, study participants and clinicians providing care to the patient in the emergency department will be blinded to the medication received.

Benefits The potential benefit of combined acetaminophen and ibuprofen therapy may provide an increased reduction in acute pain, improved patient comfort and patient/parent satisfaction compared to ibuprofen administered as a single agent. Enhanced pain reduction may potentially obviate the need for parenteral pain medication, including opioids. An additional benefit is the opportunity to contribute to research regarding pain management in children.

Risks This study may involve slightly more than minimal risk. Risk of participation in this study may be failure of combination therapy to potentiate pain reduction. Since patients will be randomized into treatment or placebo groups, they will not have the ability to choose a treatment option. Acetaminophen can be given at any age, however, there is a risk of liver toxicity in overdose. Ibuprofen has common side effects of gastrointestinal and renal effects including gastric irritation and acute renal injury. These risks, however, are considered to be minimal the medications are given as a single weight-based dose.

Data Analysis Baseline and post-treatment pain scores at 1 and 2 hours will be documented. Categorical data will be compared using the chi-squared test. Continuous data will be compared using the Mann-Whitney test for non-normally distributed data and t-test for normally distributed data. For our sample size calculation, we made the following assumptions: previous studies investigating pain scores in children have reported a decrease in pain score of 1 on a 10-point scale to be clinically significant. For this study, we assumed that a decrease in pain score of 2 would be clinically relevant. We used a standard deviation of 3 for our sample size calculation. We also assumed a 20% dropout rate and increased our sample size estimate by 15% to account for nonparametric data. Based on these assumptions, for our primary outcome, we estimated 50 patients would be needed in each group to have a power of 80% with an alpha of 0.05 to detect a difference of 2 in pain score between the two groups, with a standard deviation of 3. Data analyses of the pain scores will be based on the principle of intention to treat.

Data Safety Monitoring Plan

This is a single site study involving a biochemical intervention that presents slightly more than minimal risk due potential adverse effects from medication and randomized design. Close-monitoring will be performed by the study investigator and co-investigator every other month, or every 20 patients enrolled, whichever is more frequent. The specific procedures that will be used to monitor for and report adverse events, protocol violations and deviations are:

1. Data will be analyzed for participant recruitment
2. Data quality and protocol adherence, as determined by completeness of forms
3. Protocol adherence as determined by times of drug administration and pain assessments
4. Quality of informed consent process and documentation as determined by review of all forms for valid signatures and times
5. Analysis of adverse effects of medication determined by rates of such events as identified on data collection forms

The Data Safety Monitoring Committee Members will be:

Anthony Ciorciari, MD - Department of Emergency Medicine Michael Jones, MD - Department of Emergency Medicine Jackeline Urrutia-Monteleone, MD - Department of Pediatrics

ELIGIBILITY:
Inclusion Criteria:

* Patients with a numeric pain score of greater than or equal to 5 or Wong -Baker FACES Pain Scale of greater than or equal to 6

Exclusion Criteria:

* known allergy to ibuprofen
* Known allergy to acetaminophen
* documented or suspected pregnancy
* inability to tolerate oral medication
* a contraindication to oral intake
* inability to reliably indicate a pain score
* intake of ibuprofen or acetaminophen less than 4 hours prior to presentation
* inability to communicate in Spanish or English
* the need for immediate parenteral pain medication as per the treating physician.

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-06-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | 1 hour and 2 hours
  Change in mean pain score from baseline pain score. A validated pain score for children beginning at 3 years old, the Wong-Baker FACES pain scale (0-10 scale), will be used for patients ages 3 through 7 years. A validated numeric pain score (0-10 scale) will be used for patients 8 through 20 years. The higher score indicate worse pain.

SECONDARY OUTCOMES:
Number of participants requiring rescue medications. | 1 hour and 2 hours
  Documentation of the need for rescue medications (number and dose)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Cunningham, MD, Principal Investigator — NYCHHC - Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poddighe D, Brambilla I, Licari A, Marseglia GL. Ibuprofen for Pain Control in Children: New Value for an Old Molecule. Pediatr Emerg Care. 2019 Jun;35(6):448-453. doi: 10.1097/PEC.0000000000001505. PMID 29912084
- [Background] Gaglani A, Gross T. Pediatric Pain Management. Emerg Med Clin North Am. 2018 May;36(2):323-334. doi: 10.1016/j.emc.2017.12.002. PMID 29622325
- [Background] Jozwiak-Bebenista M, Nowak JZ. Paracetamol: mechanism of action, applications and safety concern. Acta Pol Pharm. 2014 Jan-Feb;71(1):11-23. PMID 24779190
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Gazal G, Mackie IC. A comparison of paracetamol, ibuprofen or their combination for pain relief following extractions in children under general anaesthesia: a randomized controlled trial. Int J Paediatr Dent. 2007 May;17(3):169-77. doi: 10.1111/j.1365-263X.2006.00806.x. PMID 17397460
- [Background] Motov S, Butt M, Masoudi A, Palacios W, Fassassi C, Drapkin J, Likourezos A, Hossain R, Brady J, Rothberger N, Flom P, Zerzan J, Marshall J. Comparison of Oral Ibuprofen and Acetaminophen with Either Analgesic Alone for Pediatric Emergency Department Patients with Acute Pain. J Emerg Med. 2020 May;58(5):725-732. doi: 10.1016/j.jemermed.2020.02.010. Epub 2020 Apr 1. PMID 32247660